CLINICAL TRIAL: NCT05735678
Title: Single-USe Duodenoscopes PErformance Characteristics and Technical Outcomes: the SUSPECT Italian Prospective Study
Acronym: SUSPECT
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2917
Record Dates: First submitted 2023-02-01; First posted 2023-02-21 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Disease of Gastrointestinal Tract
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Single-Use Duodenoscopes — Single-Use Duodenoscopes

SUMMARY:
Flexible endoscopes are used globally for the diagnosis and treatment of diseases of the GI tract. Duodenoscopes used for Endoscopic Retrograde Cholangiopancreatography (ERCP), in order to treat different biliary and pancreatic disorders, have been recently linked to infections transmission following the procedures. Given their reusability and their complex design of the tip with a moving metallic component, named the "elevator", these instruments must be reprocessed through high level disinfection (HLD) in order to prevent the spread of nosocomial infections. Even strict adherence to all HLD procedures results in a residual level of potentially infectious microbes. In fact, the United States Food and Drug Administration (FDA) postmarket surveillance communication reported duodenoscope culture results demonstrating contamination rates of up to 3.6% for low and moderate-concern organisms and up to 5.4% for high-concern organisms in reprocessed conventional duodenoscopes. As a consequence, at least 20 outbreaks of duodenoscope-transmitted multidrug resistant organism (MDRO) infections occurred between 2012 and 2015, despite reported compliance with duodenoscope reprocessing guidelines. The increasing concern that currents practices of reprocessing reusable duodenoscopes is insufficient, has led the FDA to released recommendation suggesting to develope a newly designed duodenoscopes. On one hand, a way is to generate duodenoscope with disposable components, such as a one-use end cap, which can be removed and allow access to the components of the elevator and other areas of the duodenoscope for reprocessing. On the other hand, an alternative is to produce a fully disposable single-use duodenoscope. The evident advantage of a single use duodenoscope, over disposable components, is that it completely eliminates the need for reprocessing and more important the risk of transmitting microbial infection from patient to patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study
* Schedule for a clinically indicated ERCP or other duodenoscope-based procedure

Exclusion Criteria:

* Potentially vulnerable subjects, including, but not limited to pregnant women
* Subjects for whom endoscopic techniques are contraindicated
* Subjects who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for a clinically indicated ERCP or other duodenoscope-based procedure will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Technical performance | 24 months
Procedural performance | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No